CLINICAL TRIAL: NCT00743587
Title: A Randomized, Double-Blind, Placebo And Active Controlled Methodology Study Investigating The Effects Of Tramadol And Naproxen On The Pain Thresholds Of Patients With Severe Pain Due To Osteoarthritis Of The Thumb
Brief Title: A Study To Assess The Ability Of Tramadol, Naproxen And Oxycodone To Affect The Pain Thresholds Of Patients With Osteoarthritis Of The Thumb
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: A9001383
Record Dates: First submitted 2008-08-28; First posted 2008-08-29 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Osteoarthritis Thumbs
MeSH Terms: interventions — Oxycodone; Tramadol; Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Placebo Comparator)
  Interventions: Drug: Placebo
- B (Active Comparator)
  Interventions: Drug: Oxycodone
- C (Active Comparator)
  Interventions: Drug: Tramadol
- D (Active Comparator)
  Interventions: Drug: Naproxen

INTERVENTIONS:
Drug: Placebo — Oral, a double-dummy approach will be used to maintain the blind between active tablet and capsule doses
  Arms: A
Drug: Oxycodone — Oral, 1 x 20mg controlled-release tablets
  Other Names: Oxycontin
  Arms: B
Drug: Tramadol — Oral, 2 x 50mg immediate release capsules
  Other Names: Dolzam
  Arms: C
Drug: Naproxen — Oral, 1 x 500mg enteric-coated
  Other Names: Naprosyne
  Arms: D

SUMMARY:
The purpose of this study is to determine if the measurement of pressure pain thresholds, in patients suffering osteoarthritis of the thumb, can be used to assess the activity of potential analgesic agents after a single dose. The study will use agents known to give pain relief in osteoarthritis as positive controls. These agents are: tramadol, naproxen and oxycodone.

ELIGIBILITY:
Inclusion Criteria:

* The clinical diagnosis of osteoarthritis of the hand, of at least 6 months duration.
* Pain around one of the thumb joints due to osteoarthritis. The patient must report the average pain in this joint, in the week prior to screening, as at least 5 on an 11-point numerical pain rating scale at the time of screening.
* The patient must demonstrate pressure pain at a thumb joint by reporting a pressure pain threshold lower than 300 kPa.

Exclusion Criteria:

* Pregnant (as judged by a urine pregnancy test) or lactating female.
* Other severe pain which may impair the assessment of the pain due to osteoarthritis.
* Skin condition over the thumb joint, which will be used for pain threshold testing, that could interfere with the assessment of pain thresholds.
* Known hypersensitivity to oxycodone, NSAIDS or tramadol.
* Patients in whom NSAIDS, oxycodone or tramadol are contraindicated, or patients taking any concurrent medications which are contraindicated with any of the study medications .
* An estimated renal clearance of less than 30 mL/min based on the Cockcroft Gault equation.
* Use of prohibited medications as listed below, in the absence of appropriate washout periods:
* Oral or intramuscular corticosteroids within 4 weeks prior to screening.
* Monoamine oxidase inhibitors within 2 weeks of screening.
* Analgesic agents, other than aspirin, or acetaminophen within 1 week prior to screening. (Aspirin use less than or equal to 325 mg per day for cardiovascular prophylaxis is permitted)
* Acetaminophen up to 4 g/day may be used, provided it is not used in the 24 hours prior to any assessment of pain thresholds.
* Intra-articular steroid injections into the study joint within 12 weeks, or to any other joint within 4 weeks, prior to screening.
* History of chronic constipation, or of any condition which, in the opinion of the investigator, may put the patient at increased risk of respiratory depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Pressure pain threshold - area under the curve | 0 to 4 hours

SECONDARY OUTCOMES:
Pressure pain threshold - at specific time points | 0 to 12 hours
Present pain intensities - at specific time points | 0 to 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9001383